CLINICAL TRIAL: NCT00597116
Title: A Randomized Phase II Trial To Evaluate The Efficacy And Safety Of Vandetanib (ZD6474, ZACTIMA ™) Versus Vinorelbine In Patients With Inoperable Or Relapsed Malignant Mesothelioma.
Brief Title: An Efficacy and Safety Study With Vandetanib to Treat Inoperable or Relapsed Malignant Mesothelioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment stopped according to early stopping rule (by protocol)
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00075; EUDRACT Number 2007-003633-16
Record Dates: First submitted 2008-01-09; First posted 2008-01-17 (Estimated); Results first posted 2012-10-15 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: Mesothelioma
Keywords: Mesothelioma; inoperable; relapsed
MeSH Terms: conditions — Mesothelioma; Recurrence | interventions — Vinorelbine; vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Vinorelbine
  Interventions: Drug: Vinorelbine
- 2 (Experimental): Vandetanib
  Interventions: Drug: Vandetanib

INTERVENTIONS:
Drug: Vinorelbine
  Other Names: Navelbine®
  Arms: 1
Drug: Vandetanib — once daily oral dose
  Other Names: ZD6474; ZACTIMA™
  Arms: 2

SUMMARY:
A clinical study to assess if a new investigational drug is effective in treating malignant mesothelioma, compared to a chemotherapy treatment (Navelbine®). In this study the patients will be assigned by chance to receive either the new drug or a chemotherapy treatment (Navelbine®). Treatment will continue as long as the cancer does not worsen and the patient wishes to continue in the study. The study will recruit approximately 66 patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mesothelioma
* Previously treated with only one course of chemotherapy for mesothelioma
* No previous treatment with vinorelbine
* No serious heart problems within the last 3 months

Exclusion Criteria:

* Serious abnormal laboratory values
* Severe or uncontrolled disease or condition as judged by the Investigator
* Pregnant or breast-feeding women
* Other cancers within the last 5 years
* Major surgery or radiation therapy within 4 weeks prior to starting study therapy
* Receipt of any investigational agents within 30 days prior to commencing study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- Germany (4):
  - Research Site, Essen
  - Research Site, Halle-Dolau
  - Research Site, Hamburg
  - Research Site, Heidelberg
- Switzerland (2):
  - Research Site, Chur
  - Research Site, Zurich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 17 December 2007, Last subject last visit: 22 July 2009.
  The study was conducted at 2 centres in Switzerland and 4 centres in Germany.
Groups:
- Vandetanib: Vandetanib 300 mg/day oral
- Vinorelbine: Vinorelbine 30 mg/m2 iv, administrated weekly
Period: Overall Study
Arm/Group | Vandetanib | Vinorelbine
Started | 14 | 11
Completed | 0 (Randomised patients ongoing study treatment at data cut-off) | 0 (Randomised patients ongoing study treatment at data cut-off)
Not Completed | 14 | 11
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Progressive disease | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib | Vinorelbine | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Median (Full Range); unit: Years] | 67 [54 to 77] | 64 [27 to 76] | 65.5 [27 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Control.
Description: Disease control is defined as having a complete response (CR), a partial response (PR) or stable disease (SD) according to the modified RECIST criteria for assessment of response in malignant pleural mesothelioma. CR is defined as the disappearance of all target lesions with no evidence of tumour elsewhere and PR is defined as at least a 30% reduction in the total tumour measurement. A confirmed response requires a repeat observation on two occasions 4 weeks apart. PD is defined as an increase of at least 20% in the total tumour measurement over the nadir measurement, or the appearance of one or more new lesions. Patients with SD are those who fulfill the criteria for neither PR nor PD.
Time Frame: Assessed at 2 months.
Population: Only patients in the evaluable for efficacy population were included.It was defined as all treated patients with no major deviations from the eligibility criteria affecting the evaluation of efficacy, who completed at least 2 cycles(unless progressive disease occurred at cycle 1)and who had at least one post-treatment tumour assessment.
Measure: Number; unit: Participants
Arm/Group | Vandetanib | Vinorelbine
Number analyzed (Participants) | 12 | 10
Participants | 0 [0 to 0] | 5 [0 to 0]

2. Secondary Outcome: Number of Participants With Objective Response.
Description: Objective response is defined as having a complete response (CR) or a partial response (PR) according to the modified RECIST criteria for assessment of response in malignant pleural mesothelioma. CR is defined as the disappearance of all target lesions with no evidence of tumour elsewhere and PR is defined as at least a 30% reduction in the total tumour measurement. A confirmed response requires a repeat observation on two occasions 4 weeks apart.
Time Frame: Assessed at 2 months.
Population: Only patients in the evaluable for efficacy population were included. It was defined as all treated patients with no major deviations from the eligibility criteria affecting the evaluation of efficacy, who completed at least 2 cycles (unless progressive disease occurred at cycle 1) and who had at least one post-treatment tumour assessment.
Measure: Number; unit: Participants
Arm/Group | Vandetanib | Vinorelbine
Number analyzed (Participants) | 12 | 10
Participants | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from randomization to date of documented response of progressive disease (PD) as assessed according to the modified RECIST criteria for assessment of response in malignant pleural mesothelioma. PD is defined as an increase of at least 20% in the total tumour measurement over the nadir measurement, or the appearance of one or more new lesions.
Time Frame: Assessed from baseline to 12 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib | Vinorelbine
Number analyzed (Participants) | 12 | 10
Months | 1.8 [1.1 to 1.8] | 3.8 [2.1 to 7.3]

4. Secondary Outcome: Overall Survival (OS)
Time Frame: Assessed from baseline to 12 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vandetanib | Vinorelbine
Number analyzed (Participants) | 12 | 10
Months | 7.8 [2.5 to 12.5] | 6.4 [3.6 to 14.9]

ADVERSE EVENTS:
Description: The enrolled and randomised population was Vandetanib 14 & Vinorelbine 11. However, demographic and baseline characteristics were analyzed for evaluable patients = safety population (Vandetanib 13 & Vinorelbine 10)
Arm/Group | Vandetanib | Vinorelbine
Serious Adverse Events (participants affected / at risk) | 6/13 | 3/10
Other Adverse Events (participants affected / at risk) | 13/13 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=13) | Vinorelbine (N=10)
Venous stasis (Vascular disorders) | 1 | 0
Acute Abdomen (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Febrile Neutropoenia (Blood and lymphatic system disorders) | 2 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Deterioration Of General Health (General disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1
Pulmonary Embolism (Vascular disorders) | 0 | 1
Papilloedema (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vandetanib (N=13) | Vinorelbine (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Ear Discomfort (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 5 | 6
Chest Pain (General disorders) | 0 | 3
General Physical Health Deterioration (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 1
Mucosal Inflammation (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 1
Orthostatic Intolerance (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3
Rhinitis (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Neutrophil Count Decreased (Infections and infestations) | 0 | 8
Weight Decreased (Infections and infestations) | 2 | 3
White Blood Cell Count Decreased (Infections and infestations) | 0 | 2
Blood Alkaline Phosphatase Increased (Infections and infestations) | 0 | 1
Liver Function Test Abnormal (Infections and infestations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 7 | 4
Diabetes Mellitus Insulin-Dependent (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 4
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Mental Disorder (Psychiatric disorders) | 1 | 0
Sleep Disorder (Psychiatric disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hot Flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.